CLINICAL TRIAL: NCT02265068
Title: Real-TICA Real Life Long-term Adherence to Ticagrelor After PCI for Acute Coronary Syndromes. Evaluation of Antiplatelet Therapy After 12 Months in Patients Undergoing PCI and Treated With Ticagrelor During the Acute Phase of an ACS.
Brief Title: Real Life Long-term Adherence to Ticagrelor After PCI for Acute Coronary Syndromes
Acronym: Real-TICA
Status: Completed | Type: Observational
Sponsor: IHF GmbH - Institut für Herzinfarktforschung (Other)
Responsible Party: Sponsor
Other Study IDs: Real-TICA
Record Dates: First submitted 2014-10-09; First posted 2014-10-15 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2017-02

CONDITIONS: Acute Coronary Syndrome (ACS)
Keywords: Acute coronary syndrome (ACS), Ticagrelor
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Ticagrelor; Dual Anti-Platelet Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ticagrelor — Treatment of ACS patients with Ticagrelor
  Other Names: Anti-platelet therapy

SUMMARY:
Documentation of long-term data regarding ticagrelor use and evaluation of reasons for discontinuation of ticagrelor in patients with ACS

DETAILED DESCRIPTION:
REAL-TICA is a retrospective non-interventional study to assess the long-term use of ticagrelor in patients with ACS and to evaluate the reasons for discontinuation of ticagrelor.

For this purpose, selected sites from the ALKK-PCI registry and the respective patients will be identified. The sites' eligibility for this study includes the frequent use of ticagrelor during the acute phase of ACS. Eligible patients are characterised by the diagnosis of ACS and the use of ticagrelor during PCI.

The eligible sites will be contacted by IHF and asked to contact their eligible patients by letter to obtain informed consent of the patients for the planned 12M follow-up by IHF. A detailed questionnaire on events within the last 12 months, current symptoms, current medication and the use of ticagrelor will be added to the patients' letters. Patients then are asked to return their responses on consent to participate in the study as well as the filled in questionnaire to IHF. Alternatively, patients may choose to receive a telephone call by IHF to answer the detailed questionnaire in person. In case of essential information missing, IHF will contact the primary care physician of the patient directly to obtain information about clinical events and medications.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* ACS (STEMI or NSTE-ACS) with PCI
* Ticagrelor treatment during the acute phase
* Written informed consent for participation in the study.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients from the ALKK-PCI registry discharged alive after PCI for ACS (STEMI and NSTE-ACS) and treated with ticagrelor during the acute phase.
Sampling Method: Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2014-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Treatment outcomes of ACS patients receiving Ticagrelor | 12 months
  Documentation of Events for ACS patients treated with Ticagrelor with follow-up over 12 months

SECONDARY OUTCOMES:
Long-term use and premature discontinuation of Ticagrelor treatment | 12 months
  Documentation of time span during which Ticagrelor is taken by patient

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Zeymer, Prof. Dr., Principal Investigator — Klinikum Ludwigshafen, Stiftung IHF - Institut für Herzinfarktforschung
Locations (6):
- Germany (6):
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Vivantes-Klinikum Neukölln, Berlin
  - Klinikum Hildesheim GmbH, Hildesheim
  - Krankenhaus Landshut-Achdorf, Landshut
  - Klinikum Ludwigshafen, Ludwigshafen
  - Klinikum-Wetzlar Braunsfeld, Wetzlar

REFERENCES:
- [Result] Zeymer U, Cully M, Hochadel M. Adherence to dual antiplatelet therapy with ticagrelor in patients with acute coronary syndromes treated with percutaneous coronary intervention in real life. Results of the REAL-TICA registry. Eur Heart J Cardiovasc Pharmacother. 2018 Oct 1;4(4):205-210. doi: 10.1093/ehjcvp/pvy018. PMID 29878086